CLINICAL TRIAL: NCT07242170
Title: Comparison of the Effectiveness of "Sciatic Nerve", "Biceps Femoris Short Head (BiFeS)" and "Interspace Between the Popliteal Artery and the Capsule of the Posterior Knee (IPACK)" Blocks Added to the Adductor Canal Block for Postoperative Pain Control in Patients Undergoing Primary Total Knee Arthroplasty: A Prospective, Randomized Controlled Clinical Trial
Brief Title: Supplementary Nerve Blocks Added to the Adductor Canal Block for Postoperative Pain Management in Primary Total Knee Arthroplasty: A Randomized Controlled Comparison of Sciatic, BiFeS, and IPACK Techniques
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, Mustafa Somunkiran, Anesthesiology resident, Erzincan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ErzincanU-ANESTEZİYOLOJİ-MS-01
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Post Operative Analgesia; Total Knee Arthroplasty
Keywords: Adductor Canal Block; Sciatic Nerve Block; Biceps Femoris Short Head Block; Interspace Between the Popliteal Artery and the Capsule of the posterior Knee block; post operative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: prospective, single-center, double-blind, randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adductor Canal Block + Sciatic Nerve Block (Experimental): Procedure: Mid-Adductor Canal Block Procedure: Sciatic Nerve Block
  Interventions: Procedure: Adductor canal block; Procedure: Sciatic Nerve Block
- Adductor Canal Block + BiFeS Block (Experimental): Procedure: Mid-Adductor Canal Block Procedure: BiFeS Block
  Interventions: Procedure: Adductor canal block; Procedure: BiFeS Block (Biceps Femoris Short Head Block)
- Adductor Canal Block + IPACK Block (Experimental): Procedure: Mid-Adductor Canal Block Procedure: IPACK Block
  Interventions: Procedure: Adductor canal block; Procedure: IPACK block

INTERVENTIONS:
Procedure: Adductor canal block — Adductor Canal Block An ultrasound-guided injection of 20 mL local anesthetic solution (10 mL 0.25% bupivacaine + 10 mL 0.9% saline) administered in the mid-portion of the adductor canal to provide motor-sparing analgesia to the anteromedial knee.
Procedure: BiFeS Block (Biceps Femoris Short Head Block) — BiFeS Block (Biceps Femoris Short Head Block) An ultrasound-guided injection targeting the short head of the biceps femoris muscle to selectively block sensory branches contributing to posterior knee pain. A total of 20 mL of local anesthetic (10 mL 0.25% bupivacaine + 10 mL 0.9% saline) is administered.
  Arms: Adductor Canal Block + BiFeS Block
Procedure: IPACK block — IPACK Block An ultrasound-guided IPACK (Interspace Between the Popliteal Artery and the Capsule of the Posterior Knee) block using 20 mL of local anesthetic solution (10 mL 0.25% bupivacaine + 10 mL 0.9% saline) to provide posterior knee capsular analgesia while sparing motor function.
  Arms: Adductor Canal Block + IPACK Block
Procedure: Sciatic Nerve Block — Sciatic Nerve Block An ultrasound-guided sciatic nerve block performed at the proximal thigh level using 20 mL of local anesthetic solution (10 mL 0.25% bupivacaine + 10 mL 0.9% saline) to provide posterior knee analgesia.
  Arms: Adductor Canal Block + Sciatic Nerve Block

SUMMARY:
Postoperative pain following total knee arthroplasty (TKA) is a significant clinical problem that delays early mobilization, reduces patient satisfaction, and increases analgesic requirements. The adductor canal block (ACB), which aims to provide analgesia while preserving motor function, is widely used in postoperative pain management after TKA. However, clinical and anatomical studies have demonstrated that ACB is effective only in the anteromedial sensory innervation of the knee and does not adequately block pain originating from the posterior knee capsule. This limitation reduces analgesic effectiveness, particularly in patients with a prominent posterior pain component.

The sciatic nerve block has long been considered the gold standard for managing posterior knee pain. However, due to disadvantages such as motor weakness and delayed rehabilitation, current pain management protocols increasingly favor motor-sparing and complementary approaches such as the Biceps Femoris Short Head (BiFeS) block and the Interspace Between the Popliteal Artery and the Capsule of the posterior Knee (IPACK) block for posterior knee analgesia.

In light of this information, the aim of our study is to guide clinical practice by comparing the postoperative analgesic efficacy, motor function outcomes, and patient satisfaction associated with sciatic nerve, BiFeS, and IPACK block techniques-each administered as a supplement to the adductor canal block-in patients undergoing total knee arthroplasty, with the ultimate goal of determining the optimal block combination for postoperative pain control.

DETAILED DESCRIPTION:
The study was designed as a prospective, single-center, double-blind, randomized controlled trial to be conducted in the operating rooms of Erzincan Binali Yıldırım University Mengücek Gazi Training and Research Hospital. The study will begin after obtaining approval from the Erzincan Binali Yıldırım University Ethics Committee and written informed consent from all participants. A minimum of 102 patients (based on G-Power analysis), aged 18-75 years, scheduled for elective unilateral primary total knee arthroplasty by the Orthopedics and Traumatology Department and classified as American Society of Anesthesiologists (ASA) physical status I-III, will be included.

Patients with ASA ≥ IV, those undergoing revision total knee arthroplasty, bilateral arthroplasty, neuromuscular disease, cognitive dysfunction, drug allergies, a history of local anesthetic systemic toxicity, neurological deficits, bleeding diathesis, pregnancy, or those who decline participation will be excluded. The study will be conducted over a 12-month period between November 1, 2025 and November 1, 2026.

All patients will be informed about the study protocol and procedures one day before surgery, and written consent will be obtained. Upon arrival to the operating room, standard monitoring will be applied. As per routine practice, spinal anesthesia will be performed. Nasal oxygen at 2 L/min will be administered. During surgery, standard hemodynamic parameters (SpO₂, blood pressure, heart rate) will be recorded.

Spinal anesthesia will be conducted according to standard regional anesthesia protocols for total knee arthroplasty using a 25-gauge pencil-point spinal needle at the L3-L4 interspace in the sitting position. A total of 15 mg (3 mL) of 0.5% hyperbaric bupivacaine and 20 mcg (0.4 mL) fentanyl will be administered. Surgery will commence once a T10 sensory block level is achieved. Motor block will be assessed using the Modified Bromage Scale, and sensory block using pinprick or cold tests to determine dermatomal level.

At the end of surgery, under sterile conditions and ultrasound (USG) guidance, patients assigned to Group I will receive a Mid-Adductor Canal block with 20 mL (10 mL 0.25% bupivacaine + 10 mL 0.9% NaCl) and a Sciatic nerve block with 20 mL of the same local anesthetic solution. Group II patients will receive a Mid-Adductor Canal block and a BiFeS (Biceps Femoris Short Head) block using identical volumes and concentrations. Group III patients will receive a Mid-Adductor Canal block and an IPACK (Interspace Between the Popliteal Artery and the Capsule of the Posterior Knee) block with the same solution. All blocks will be performed by a single anesthesiologist with at least 3 years of experience in peripheral nerve blocks. Anesthesia technicians, operating room nurses, and postoperative assessors will be blinded to group allocation.

Patients will be randomized in a 1:1:1 ratio into three groups (Group I: Mid-Adductor Canal + Sciatic; Group II: Mid-Adductor Canal + BiFeS; Group III: Mid-Adductor Canal + IPACK). The randomization sequence was generated by a blinded statistician using computer-generated permuted blocks (block size = 6). To minimize prognostic imbalance, stratification was performed according to body mass index (BMI <30 / ≥30) and age (<66 / ≥66). Separate permuted block lists were created for each stratum, yielding: S1 (BMI<30, <66): 26; S2 (BMI<30, ≥66): 25; S3 (BMI≥30, <66): 26; S4 (BMI≥30, ≥66): 25 envelopes. Full blocks achieved a 1:1:1 balance within each stratum; partial blocks were algorithmically assigned to maintain stratified balance. Equal distribution across groups (34/34/34) was targeted.

Allocation concealment was ensured using sequentially numbered, opaque, sealed envelopes (SNOSE) prepared separately for each stratum by an investigator blinded to group assignments. Envelopes were stored in a locked cabinet. For each eligible patient, the anesthesiologist performing the intervention opened the next envelope corresponding to that patient's stratum at the end of surgery. While the anesthesiologist performing the block was aware of the allocation, postoperative data collectors and outcome assessors remained blinded. Randomization lists remained inaccessible until completion of data collection and were unblinded only during analysis.

After the procedure, patients will be transferred to the postoperative care unit as per routine. When the Aldrete score reaches ≥9, patients will be transferred to the ward. All patients will receive standard multimodal analgesia including IV paracetamol 1 g every 8 hours, IV ibuprofen 400 mg every 12 hours, and intravenous tramadol hydrochloride is planned to be used as rescue analgesia (rescue opioid) when needed. Tramadol hydrochloride administration will be regulated at a dose of 100 mg IV (intravenous), limited to a maximum of 400 mg (4 doses) within 24 hours.

VAS scores will be recorded at postoperative hours 1, 4, 8, 12, and 24. Motor block will be evaluated using the Modified Bromage Scale and peroneal nerve motor function via ankle dorsiflexion and great toe extension tests. Rescue opioid usage and time to first opioid requirement will be documented during the first 24 hours. All patients will complete the Quality of Recovery-40 (QoR-40) questionnaire at postoperative hour 24. Postoperative evaluations will be performed by a physician blinded to the type of block. PACU and ward nurses will also remain blinded to group assignments.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified as American Society of Anesthesiologists (ASA) physical status I-III
* Patients undergoing primary total knee arthroplasty
* Patients undergoing unilateral total knee arthroplasty
* Patients between 18 and 75 years of age

Exclusion Criteria:

* Patients classified as American Society of Anesthesiologists (ASA) physical status IV or higher
* Patients undergoing revision total knee arthroplasty
* Patients undergoing bilateral total knee arthroplasty
* Patients with neuromuscular disease
* Patients who decline to participate in the study
* Patients with cognitive dysfunction
* Patients with known drug allergies
* Patients with a history of local anesthetic systemic toxicity
* Patients with neurological dysfunction
* Patients with bleeding diathesis
* Pregnant patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Pain Score | Postoperative 24 hours (measured at 1, 4, 8, 12, and 24 hours)
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a 10-cm horizontal line with endpoints representing the extremes of pain (0 = "no pain," 10 = "worst imaginable pain"). Patients will mark their perceived pain level, and the distance (in cm or mm) from the "no pain" anchor will be recorded as the VAS score. Measurements will be performed at rest. A VAS score below 3 indicates mild pain and adequate analgesia.

SECONDARY OUTCOMES:
Modified Bromage Scale | 24 hours
  The Modified Bromage Scale is widely used to objectively assess the degree of motor block following spinal or peripheral nerve blocks. The evaluation will be performed after the resolution of spinal anesthesia and during the postoperative period while the peripheral nerve block remains effective.
  The scores obtained will be recorded to determine the degree of motor block and its potential effects on early mobilization.
  Score 0 - The patient can freely move the lower extremity (hip, knee, ankle). Score 1 - The patient can move the knee and ankle but cannot move the hip. Score 2 - The patient can move only the ankle; unable to move the knee and hip. Score 3 - The patient is unable to move the lower extremity at all.
QoR-40 (Quality of Recovery-40) Questionnaire | 24 hours
  The QoR-40 is a validated and reliable multidimensional instrument designed to assess postoperative recovery. The questionnaire consists of 40 items, each scored on a 5-point Likert scale:
  1: Strongly disagree / very poor
  5: Strongly agree / excellent
  Total scores range from 40 to 200, with higher scores indicating better quality of recovery.
  The QoR-40 evaluates five subdomains:
  Physical comfort (12 items)
  Emotional state (9 items)
  Physical independence (5 items)
  Psychological support (7 items)
  Pain (7 items)
  All patients will complete the questionnaire at the postoperative 24th hour, after receiving verbal instructions. The resulting scores will be analyzed to compare the effects of each block combination on patient comfort and overall recovery quality.
Postoperative Opioid Requirement | 24 hours
  The amount of opioid analgesics required during the postoperative period.
Time to First Opioid Requirement | 24 hours
  The time to first opioid requirement will be assessed by recording the time the patient requests or receives their first opioid dose post-operatively.
Peroneal nerve motor function | 24 hours
  Peroneal nerve motor function will be assessed using ankle dorsiflexion and great toe extension tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan Binali Yıldırım Üniversitesi, Erzincan, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No